CLINICAL TRIAL: NCT02356055
Title: High-dose Mass Practice Intervention to Reduce ADL Disability in Dementia
Brief Title: Mass Practice of Activities of Daily Living in Dementia (STOMP)
Acronym: STOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); OU Medical Center (Unknown); Oklahoma Shared Clinical and Translational Resources (Other); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4648
Record Dates: First submitted 2014-10-07; First posted 2015-02-05 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: activities of daily living; massed practice; occupational therapy
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Protocol (Experimental): Participants in this group will receive the Skill-building through Task-Oriented Motor Practice (STOMP) intervention 3 hours/day, 5 days/week for 2 weeks. Participants will choose functional goals that have an identifiable beginning and concluding step for creation of "practice-able" steps for task-oriented training. Practice-able steps will embed both task modifications and assistive technology determined by the OT to support performance and will be situated contextually within the participant's habits and environment. Each group will practice the task as many times as possible during their allotted time in training. For the intensive protocol, each hour of training will focus on 1 of 3 identified goals and will include 50 minutes of intervention and a 10 minute break.
  Interventions: Behavioral: STOMP (Skill-building through Task-Oriented Motor Practice)
- Less-Intensive Protocol (Active Comparator): Participants in this group will receive the Skill-building through Task-Oriented Motor Practice (STOMP) intervention 1 hour/day, 2 days/week for 2 weeks. Participants will choose goals that have an identifiable beginning and concluding step for creation of "practice-able" steps for task-oriented training. Practice-able steps will embed both task modifications and assistive technology determined by the OT to support performance and will be situated contextually within the participant's habits and environment. Each group will practice the task as many times as possible during their allotted time in training. In the less-intensive protocol, each of the 3 ADL goals will be practiced as many times as possible within 20 minutes of the scheduled hour.
  Interventions: Behavioral: STOMP (Skill-building through Task-Oriented Motor Practice)

INTERVENTIONS:
Behavioral: STOMP (Skill-building through Task-Oriented Motor Practice) — The STOMP intervention is a package including family-centered goals, task-specific training delivered through motor learning and errorless learning principles. It is unique in the use of massed practice (high-dosage) therapy.

SUMMARY:
People with Alzheimer's disease and related dementias present with changes in how they think, move and emotionally respond to daily life situations. While type of dementia will dictate how severe certain symptoms are, all people with dementia will report a gradual change in how they function in daily life skills. Losing the ability to do daily life tasks, such as using a cell phone, balance a checkbook or get dressed in the morning signifies loss for both the person with dementia and their caregiver. Caregivers that assist with daily life tasks report more depression and anxiety, as well as a higher burden of care. People with dementia that lose the ability to perform daily tasks report more depression and decreased satisfaction with life. Despite gains in research, researchers are still missing important pieces that will improve rehabilitation interventions for improving daily life skills.

In order to address the needs of people with dementia, an intervention called Skill-building through Task-Oriented Motor Practice (STOMP) was developed by an occupational therapist. Our team proposes that improvement in daily life skills is possible under certain circumstances. First, the daily life task a person is addressing in rehabilitation should be personally-meaningful and should also be the task practiced in therapy which is called "task-oriented training". For example, a person that is having trouble making a sandwich should practice making a sandwich. Second, the investigators propose that people with dementia need a lot of "correct practice" so that the brain has time to "rewire" how to do the task correctly. Therefore, when patients practice tasks using STOMP, investigators do not allow our participants to make errors and patients practice for long periods of time. Investigators also incorporate and provide new technology into training such as medication reminder alarms and photo phones which allow you to dial a number by choosing a loved one's picture.

In this pilot study, the investigators want to look more closely at the how the amount of time you practice influences study outcomes. The investigators believe that the findings from this study will support our belief that more time in therapy is needed to enhance how someone with dementia learns.

DETAILED DESCRIPTION:
A. BACKGROUND: Progressive disability in activities of daily living (ADL) is inevitable for people with Alzheimer's disease and related dementias (ADRD). Attempts to slow or prevent ADL disability have been unsuccessful despite making progress in behavioral training methods. Missing from this research is an emphasis on how investigators maximize a patient's engagement during training and the rigorous examination of implementation protocols (dosing and training methods) which may advantage learning in people with ADRD. Our team addressed this gap with the development of the STOMP (Skill-building through Task-Oriented Motor Practice) intervention which creates methods for obtaining ADL goals that support "personhood" and tests high-intensity protocols that appear to advantage learning as well as sustained learning over time. Through our first specific aim, the investigators will examine the learning and retention of learning advantages offered through receipt of an intensive versus less-intensive STOMP protocol. In our second aim,the investigators will examine sustained attention to task during training as a differential contributor to our outcomes.

B. RESEARCH DESIGN/METHODS

1. Design: Randomized-controlled trial over a two-week intervention period and a 3-month post-intervention follow-up period that will occur over 24 months. The investigators will employ block randomization where participants are randomized in blocks of randomly chosen sets of two or four, ultimately resulting in eight participants randomized to each group in the first year and a total of 16 participants assigned to each group by the end of 20 months. Two occupational therapists (OT), blinded to group assignment will complete baseline, post-intervention and 3-month follow-up assessments. The treating occupational therapy assistant (OTA) will be given the group assignment by the PI after the baseline evaluation is complete.
2. Recruitment: The investigators intend to recruit 32 participants (through assent) and legally-authorized representatives (through informed consent) employing a variety of methods. The primary recruitment strategy will be the use of direct mailing which has been successfully used by other teams recruiting people with ADRD.9 A letter of invitation explaining the study and ways to participate will be mailed to zip codes adjacent to University of Oklahoma Health Sciences Center (OUHSC) through the United States Postal Service. Second, collaborating physicians (Drs. Hershey and Odenheimer) will refer appropriate candidates. Dr. Hershey, a neurologist specializing in dementia diagnosis and treatment with OUHSC, sees >200 people/year with various forms of dementia. Dr. Odenheimer, a neurologist with the VA sees 30 new patients/year with dementia and 45 unique return visits/year. Other forms of recruitment will include: media (e.g., campus emails, newspaper advertisements, websites, television news stories) and presentations at local chapters of the Alzheimer's Association support group. Previous recruitment has occurred primarily through media/presentations (60%) and physician recruitment (40%).
3. Procedures: Figure 2 clearly outlines the manualized study procedures which are taught to the OT/OTA through a 40-hour certification course. Protocol preparation: The Canadian Occupational Performance Measure (COPM) includes a semi-structured interview that will assist the OT in facilitating family/participant chosen ADL, home management or leisure goals that support retention of personhood for the person with dementia. Goals chosen through the COPM are performed by the participant and assessed by the OT in order to develop measurable GAS outcomes. Each goal must have an identifiable beginning and concluding step for creation of "practice-able" steps for task-oriented training. Practice-able steps will embed both task modifications and assistive technology determined by the OT to support performance and will be situated contextually within the participant's habits and environment. To enhance transfer of training to the caregivers, we will invite caregivers to watch the intervention daily and require hands-on training of the intervention one day/week. The intervention protocol incorporates important multi-component features of motor learning. Each group will practice the task as many times as possible during their allotted time in training. For the intensive protocol, each hour of training will focus on 1 of 3 identified goals and will include 50 minutes of intervention and a 10 minute break. The less-intensive protocol is based on home health treatment protocols where patients are seen 1-2 days/week for one hour/day. In the less-intensive protocol, each of the 3 ADL goals will be practiced as many times as possible within 20 minutes of the scheduled hour. In both protocols, the OTA will employ errorless learning where the participant is prevented from making errors through scaffolded trainer guidance progressing from hand-over-hand training, provision of tactile and verbal cues and, if possible, no cues for errorless performance. Continuous verbal feedback will be provided to the participant initially and minimized as training progresses. Post-intervention, caregiver support for questions and problems interfering with continued practice is provided monthly until the 3-month follow-up.
4. Statistical Methods A two-sided 0.05 alpha level will be used to define statistical significance. An intent-to-treat paradigm will be followed in which data from all randomized patients are analyzed to intervention assignment without regard to adherence or outcomes.

   Aim 1: Examine advantages to learning and retention of learning provided through receipt of the intensive STOMP protocol versus a less-intensive protocol.

   Plan: Changes in pre- and post-intervention (immediate and 90 day) GAS T-scores/COPM mean scores will be compared between intervention groups using a repeated measures ANOVA where time by intervention interaction term will be tested to determine if the estimated effect of the intervention program differs over the follow-up period. Analyses will be stratified by post-intervention time point if a significant interaction is found. Residual diagnostics will be created to assess adequacy of modeling assumptions. Non-parametric analyses will be used, focusing on 3-month differences, if ANOVA modeling assumptions are not satisfied.

   Aim 2: Examine sustained attention to task as a contributor to differential outcomes.

   Plan: Using data from the Sustained Attention to Task behavioral form (Sec.3f), we will tally the amount of time spent on each of 3 ADL goals over the 2 week intervention. Total minutes on task will be categorized by tertiles and plotted against change in GAS and COPM scores, both post-intervention and the 3-month follow-up.
5. Study Timeline*

   * Patient follow-up completed by month 23 to assure time for final data analysis.
6. Data Management: Data capture, quality assurance, management, and processing will be consolidated through the use of the well-established Research Electronic Data Capture (REDCap) system.10 REDCap is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources. Online data capture forms will be created using REDCap, exported as pdf files, and printed for off-line use so that a hard copy will be available for data checks. REDCap will allow for multi-personnel access of project files and will be used by the PI, evaluators and trainer to capture data.

C. POTENTIAL PROBLEMS AND ALTERNATIVE APPROACHES Three hours of intervention daily may result in fatigue, refusals and displays of negative behaviors. Due to the repetitive nature of STOMP, we have tallied the number of negative behaviors to include wandering, purposeless movement, verbal and physical outburst and mood-related verbalizations and have averaged <1/hour across 3 hours of treatment in both settings.1,2 We believe this success is in part due to 1) using licensed OT/OTAs; 2) training the interventionists through a manualized, STOMP protocol which includes the identification of behavioral signs with specific redirections for negative behaviors; and 3) engaging the presence of the caregiver. Recruitment for our home-based studies has proven to be more palatable to community-dwelling older adults than clinic-based. Based on our previous work, we believe that the 30 day phone calls have largely influenced our ability to retain 100% of our participants at 90-day post-intervention follow-up.

D. HUMAN PARTICIPANT SAFETY The risk for participating in this study is similar to doing ADL tasks at home. Strict safety principles will be observed such as walking with a safety belt as deemed necessary. The benefits of participating in the study include assessment of deficits with an occupational therapist, receiving two weeks of free intervention, and provision of adaptive equipment that will support functional skills in the home. The investigators believe the benefits of participating outweigh the risks.

ELIGIBILITY:
Inclusion Criteria:

1. Lives in the community and speaks English
2. adult aged 50-90 years old
3. lives with someone who can provide consent to be in the study
4. diagnosed with some form of dementia
5. cognitive score on the Mini-Mental Status Examination score >10 but ≤25
6. able to understand and follow one step commands
7. can move one arm sufficiently for practicing tasks
8. participant or family member can identify three goal areas related to self-care or home management
9. able to participate in 3 hours of daily therapy in their home environment for 2 consecutive weeks

Exclusion Criteria:

1. Creutzfeldt-Jakob Dementia, delirium or a progressive neurological condition such as Parkinson's disease
2. receptive or global aphasia
3. uncorrected vision/hearing

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
5 point Observation of Activities of Daily Living | Baseline
  The investigator observes ADL and then using an ordinal measure (-2, -1, 0, 1, 2), the
  researcher breaks the patient goal into five possible scenarios where "0" equals the intended goal (determined after researcher observation); negative scores represent "much less" and "somewhat less" than the expected outcome and positive scores represent "somewhat more" and "much more" than expected outcome.

SECONDARY OUTCOMES:
Frequency of Behavioral Responses during the Trial | Daily for 2 weeks
  Sustained attention to task" is recorded during each intervention using a stopwatch. When a participant stops practicing the task for any reason and does not return to task within 30 seconds, the stopwatch is stopped and sustained attention for each unit of engaged time is recorded. In the end, the episodes of time on task for each day are tallied. "Number of repetitions" is recorded as repetitions occur and tallied to represent the number of repetitions completed for each task in each hour. Neuropsychiatric behaviors, such as verbal and physical aggression, are recorded as they occur on a 3rd behavior tracking form.
10 point Caregiver Perception of Activity of Daily Living Performance and Satisfaction with Performance | Baseline
  The caregiver or client identifies tasks that are most important and then reports performance and satisfaction with performance on each task on a scale of 1-10 (1=worst, 10=best).
Change in 10 point Caregiver Perception of Activity of Daily Living Performance and Satisfaction with Performance | Post-intervention (within 72 hours)
  The caregiver reports performance and satisfaction with performance on each task on a scale of 1-10 (1=worst, 10=best).
Retention of 10 point Caregiver Perception of Activity of Daily Living Performance and Satisfaction with Performance | 90 days
  The caregiver reports performance and satisfaction with performance on each task on a scale of 1-10 (1=worst, 10=best).
Change in Observation of Activity of Daily Living | Post-intervention (within 72 hours)
  Status of observed Activity of daily living after intervention within 72 hours
Retention of Observed Activity of Daily Living at 90 Days | 90 days
  Status of observed ADL using 5 point scale 90 days after the intervention is over

CONTACTS AND LOCATIONS:
Overall Officials: Carrie A Ciro, PhD, OTR/L, Principal Investigator — University of Oklahoma

REFERENCES:
- [Derived] Ciro CA, Stoner J, Prodan C, Hershey L. Skill-building through Task-Oriented Motor Practice (STOMP) intervention for activities of daily living: study protocol for a randomized, single blinded clinical trial. Clin Trials Degener Dis. 2016 Apr-Jun;1(2):45-50. doi: 10.4103/2468-5658.184743. Epub 2016 Jul 7. PMID 29071307